CLINICAL TRIAL: NCT02743377
Title: PET Imaging of Phosphodiesterase-4 (PDE4) in Brain and Peripheral Organs of Mccune-Albright Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 160093; 16-M-0093
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-05-19

CONDITIONS: Nervous System Disease
Keywords: GsI+/-; Camp; GNAS
MeSH Terms: conditions — Nervous System Diseases; Muscle Cramp | interventions — Roflumilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with McCune-Albright syndrome (MAS) (Experimental): Subjects with McCune-Albright syndrome (MAS) who received 11C-(R)-rolipram whole-body and/or brain PET scans
  Interventions: Other: Brain PET Imaging with 11C Rolipram; Drug: Whole Body PET Baseline with 11C Rolipram; Drug: Whole Body PET Blocked with Roflumilast
- Healthy control (Experimental): Healthy control received 11C-(R)-rolipram whole-body and/or brain PET scans
  Interventions: Other: Brain PET Imaging with 11C Rolipram; Drug: Whole Body PET Baseline with 11C Rolipram

INTERVENTIONS:
Other: Brain PET Imaging with 11C Rolipram — Brain PET Imaging, single scan, with 11C Rolipram 20 mCi given intravenously at the start of the scan
Drug: Whole Body PET Baseline with 11C Rolipram — Whole Body Baseline PET Imaging, single scan, with 11C Rolipram 20 mCi given intravenously at the start of the scan
Drug: Whole Body PET Blocked with Roflumilast — Whole Body PET Imaging scan after blockade with Roflumilast 500 mcg PO, given 1-2 hours prior to start of scan
  Arms: Subjects with McCune-Albright syndrome (MAS)

SUMMARY:
Background:

McCune-Albright Syndrome (MAS) is a disorder that affects the bones, skin, and some hormone-producing tissues. It is associated with a mutation in a gene. This gene affects enzymes in the brain and body. Researchers want to learn more about one of these enzymes, Phosphodiesterase 4 (PDE4), in people with MAS.

Objective:

To see if people with MAS have higher levels of PDE4 than people without MAS.

Eligibility:

People ages 18 and older who have MAS and participated in protocol 98-D-0145, Screening and Natural History of Patients with Polyostotic Fibrous Dysplasia and the McCune-Albright Syndrome. Healthy adult volunteers are also needed.

Design:

This study requires 1 to 4 outpatient visits to the NIH Clinical Center. Some visits may take place on the same day.

Participants with MAS will be screened with medical history and physical exam. They will have blood and urine tests.

Participants will have a magnetic resonance imaging scan.

Participants will have a full body positron emission tomography (PET) scan. A small amount of a radioactive chemical, [11C](R)-rolipram, will be given through an intravenous tube.

Participants will have a brain PET scan with [11C](R)-rolipram. For this, a thin plastic tube will also be put into an artery at their wrist or elbow crease area.

For the scans, participants will lie on a bed that slides in and out of a scanner. They may wear a plastic mask to hold their head in place. They will have blood drawn.

Participants with MAS will be interviewed about their thinking and mood. They may complete questionnaires about how they feel or think.

DETAILED DESCRIPTION:
Objective: McCune-Albright syndrome (MAS) is a mosaic disease arising from early embryonic somatic activating mutations of GNAS, which encodes the 3 <=, 5 <=-cyclic adenosine monophosphate (cAMP) pathway-associated G-protein, Gs . Constitutive activation of Gs leads to increased cAMP signaling in brain, as well as in peripheral organs, particularly bones. Although subjects with MAS show psychiatric and neurological symptoms, few studies have attempted to assess brain changes in these individuals. This protocol seeks to study changes in the cAMP cascade both in brain and peripheral organs of individuals with MAS using [11C](R)-rolipram PET, which binds to phosphodiesterase 4 (PDE4) and reflects cAMP cascade activity.

Study population: Participants will include 20 subjects with MAS and 15 healthy subjects group-matched to MAS subjects for age and gender. Both MAS subjects and healthy controls will have one or two PET scans: one whole body and one brain scan. We expect about 10 brain and 10 whole body scan to be performed in each group.

Design: Subjects with MAS will be recruited from participants in 98-D-0145 Screening and Natural History of Patients with Polyostotic Fibrous Dysplasia and the McCune-Albright Syndrome (PI: Alison M. Boyce, MD). Only participants in protocol (98-D-0145) who provided self-consent without a legally authorized representative will be recruited. Brain PET scans will be performed by measuring metabolite-corrected arterial input function. No venous blood sampling will be performed for whole body scans.

Outcome measures: The primary outcome measure will be obtained in brain scans as the amount of radioligand binding quantified as distribution volume (Vt). Calculated from both brain and plasma data, Vt reflects rolipram binding to PDE4, corrected for any individual differences in metabolism of the radioligand or regional blood flow in brain. The secondary outcome measure will be obtained in whole body scans as area under the curve (AUC) of radioactivity expressed as standard uptake value (SUV). SUV is calculated by normalizing radioactivity in PET images to injection activity and body weight. Vt in brain will be compared between subjects with MAS and healthy controls. AUC will be compared within-subjects with MAS between areas of craniofacial fibrous dysplasia and adjacent unaffected bone. AUC of whole body scans will also be compared between subjects with MAS and healthy controls. We hypothesize that subjects with MAS will show greater rolipram binding than healthy controls in brain regions, as well as greater rolipram uptake in bones affected by fibrous dysplasia than in unaffected bones.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with MAS:

* At least 18 years of age
* Able to provide self-consent
* Diagnosed with MAS under 98-D-0145.
* Have craniofacial fibrous dysplasia

Healthy Subjects:

* At least 18 years of age.
* Healthy based on medical history and physical examination.

EXCLUSION CRITERIA:

Subjects with MAS:

* Serious medical conditions, which may interfere with study procedures. Such conditions include but not limited to significant bone abnormalities in wrist areas of both arms, which makes it difficult to place a radial arterial line, clinically marked dysfunction of liver or kidney, which may delay clearance of [(11)C](R)-rolipram.
* Clinically significant laboratory abnormalities not linked to endocrine abnormalities but that may interfere with the PET measurement or affect safety of the participant during this study.
* Positive HIV test.
* Head trauma resulting in a period of unconsciousness lasting longer than one hour.
* Metallic foreign bodies that would be affected by the magnetic resonance imaging (MRI) magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
* Recent research-related exposure to radiation (i.e., PET from other research) that, when combined with this study, would be above the allowable limits.
* Inability to lie flat on camera bed for about two and a half hours.
* Pregnancy or breastfeeding.
* NIMH employees/staff and their immediate family members will be excluded from the study per NIMH policy.

Healthy Subjects:

* Serious medical conditions, which may interfere with study procedures. Such conditions include but not limited to clinically marked dysfunction of liver or kidney, which may delay clearance of [(11)C](R)-rolipram.
* Clinically significant laboratory abnormalities that may interfere with the PET measurement or affect safety of the participant during this study.
* Personal history of any DSM Axis I disorder.
* Positive HIV test.
* Head trauma resulting in a period of unconsciousness lasting longer than one hour.
* Metallic foreign bodies that would be affected by the MRI magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
* Recent research-related exposure to radiation (i.e., PET from other research) that, when combined with this study, would be above the allowable limits.
* Inability to lie flat on camera bed for about two and a half hours.
* Pregnancy or breastfeeding.
* Current substance use disorder based on DSM.
* NIMH employees/staff and their immediate family members will be excluded from the study per NIMH policy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-M-0093.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 subjects were enrolled but one subject did not start the study.
Groups:
- Healthy Control: Healthy controls received 11C-(R)-rolipram whole-body and/or brain PET scans
Period: Overall Study
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Started | 9 | 6
Brain PET With 11C Rolipram | 8 | 3
Whole Body PET Baseline With 11C Rolipra | 5 | 4
Whole Body PET Baseline & Blocked | 0 | 2
Completed | 7 | 6
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS) | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (30-120min) - Bladder
Description: Determine if there is a difference in PDE4 levels (measured using [11C]rolipram) in the periphery of patients with McCune-Albright Syndrome (MAS) compared to healthy controls.
Time Frame: 120 minutes
Population: Subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 5 | 4
SUV x min | 575.1 (402.2) | 650.8 (344.7)

2. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (30-120min) -Gallbladder
Description: as for outcome 1
Time Frame: 120 minutes
Population: Subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 5 | 4
SUV x min | 581.2 (235.8) | 417.9 (317.8)

3. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (30-120min) - Heart
Description: as for outcome 1
Time Frame: 120 minutes
Population: Subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 5 | 4
SUV x min | 27.4 (6.1) | 25.4 (5.8)

4. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (30-120min) - Kidneys
Description: as for outcome 1
Time Frame: 120 minutes
Population: Subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 5 | 4
SUV x min | 63.3 (14.8) | 80.4 (12.4)

5. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (30-120min) - Liver
Description: as for outcome 1
Time Frame: 120 minutes
Population: Subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 5 | 4
SUV x min | 47.6 (21.7) | 52.4 (4.4)

6. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (30-120min) - Lungs
Description: as for outcome 1
Time Frame: 120 minutes
Population: Subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 5 | 4
SUV x min | 10.2 (4.3) | 9.6 (4.4)

7. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (30-120min) -Spleen
Description: as for outcome 1
Time Frame: 120 minutes
Population: Subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 5 | 4
SUV x min | 20.1 (2.8) | 18.7 (2.7)

8. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (30-120min) - Stomach
Description: as for outcome 1
Time Frame: 120 minutes
Population: Subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 5 | 4
SUV x min | 39.4 (20.8) | 34.1 (22.8)

9. Primary Outcome: Whole Brain Total Distribution Volume (VT)
Description: Determine if there is a difference in PDE4 levels (measured using [11C]rolipram) in the brain of patients with McCune-Albright Syndrome (MAS) compared to healthy controls
Time Frame: 90 minutes
Population: Subjects who completed brain scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: mL x cm-3
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 7 | 3
mL x cm-3 | 0.67 (0.08) | 0.52 (0.06)

10. Primary Outcome: MAS Affected Bone SUV AUC(60-120min) at Baseline
Description: To assess whether uptake in dysplastic bone reflects parent radioligand binding to the enzyme or merely accumulation of radiometabolites
Time Frame: 120 minutes
Population: Subjects who completed two whole body scans the first with 11-C Rolipram, and the second blocked with Roflumilast
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 2
SUV x min | 11.2 (0.66)

11. Primary Outcome: MAS Affected Bone SUV AUC(60-120min) - Blocked
Description: as for outcome 10
Time Frame: 120 minutes
Population: Subjects who completed two whole body scans, the first with 11-C Rolipram and the second blocked with Roflumilast
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 2
SUV x min | 11.1 (0.53)

12. Secondary Outcome: MAS Affected Bone SUV AUC(60-120min) - for Baseline and Blocked Subjects With MAS
Description: Determine if PDE4 levels are different in areas of fibrous dysplasia as compared to unaffected bones in patients with MAS
Time Frame: 120 minutes
Population: The analyses included two group of subjects with MAS: subjects who completed a whole body PET scan with 11-C Rolipram and subjects who completed whole body PET scan after blockade with Roflumilast 500 mcg PO
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Subjects With McCune-Albright Syndrome (MAS)
Number analyzed (Participants) | 6
SUV x min | 13.5 (2)

13. Secondary Outcome: Normal Bone SUV AUC (60-120min) - for Healthy Controls
Description: as for outcome 12
Time Frame: 120 minutes after the start of the scan
Population: Healthy control subjects who completed whole body scan with 11-C Rolipram
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Healthy Control
Number analyzed (Participants) | 5
SUV x min | 4.2 (3.4)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Subjects With McCune-Albright Syndrome (MAS): Subjects with McCune-Albright syndrome (MAS) received 11C-(R)-rolipram whole-body and/or brain PET scans
Arm/Group | Healthy Control | Subjects With McCune-Albright Syndrome (MAS)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 3/9 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Control (N=9) | Subjects With McCune-Albright Syndrome (MAS) (N=6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02743377/Prot_SAP_000.pdf